CLINICAL TRIAL: NCT03443128
Title: Phase II Study of Vinorelbine for Children with Recurrent Anaplastic Large Cell Lymphoma
Brief Title: Vinorelbine for Recurrent ALCL-2017
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Cancer Group, China (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCGChina-R-ALCL-2017
Record Dates: First submitted 2018-02-17; First posted 2018-02-22 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Anaplastic Large Cell Lymphoma; Vinorelbine
Keywords: Anaplastic Large Cell Lymphoma; Recurrent; Childhood; Adolescent; Treatment
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic; Recurrence | interventions — Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vinorelbine monotherapy treatment (Experimental): Patients will be treated with Vinorelbine. Four weeks as a course. There are 20 courses in total.
  Interventions: Drug: Vinorelbine

INTERVENTIONS:
Drug: Vinorelbine — During each course, patients will be treated with vinorelbine (25mg/m2/week on weeks 1-3). After 1 course(4 weeks) of vinorelbine, response will be evaluated by simple assessment: clinical symptoms, signs, B ultrasound, chest X-ray, peripheral blood test and bone marrow smear(if needed). After 2 courses, response will be evaluatedy by simple assessment, CT and FDG-PET. The CR/CRu was defined by anatomic tumour shrinkage more than 75% after 2 courses based on CT with negative PET assessment, with negative bone marrow PCR(if needed) and without CNS involvement. Patients who achieved a CR/CRu after two courses either will proceed to stem cell transplantation (SCT) or will receive additional courses of therapy while awaiting SCT. Response was re-evaluated at the end of every 2 courses. Patients with progressive disease at any time during treatment will be removed from protocol therapy.

SUMMARY:
The purpose of this study is to assess the efficiency and safety of vinorelbine in the treatment of relapsed / advanced ALCL in children and adolescents.

DETAILED DESCRIPTION:
Anaplastic large cell lymphoma (ALCL) is a rare non-Hodgkin's lymphoma, around 30% patients would get relapse. Vinorelbine(Navelbine) is a third-line treatment option for Hodgkin's disease(HD) after transplantation failed, while both HD and ALCL express CD30. When ALCL recurred, vinblastine monotherapy was used and the 5-year EFS up to 30%, 5-year OS up to 60%. In China vinblastine is unavailable. Vinorelbine is very similar to vinblastine in molecular formula, and is available in China. From November 2016 to March 2017, two patients with recurrent ALCL were recruited in the Department of Hematology and Oncology, Shanghai Children's Medical Center. They received vinorelbine monotherapy and achieved clinical remission (PET CR) at 8 weeks. One patient with bone marrow recurrence showed negative ALK / NPM by PCR . Based on this, the investigators will expand the sample to further investigate the therapeutic efficiency and safety of vinorelbine in children and adolescents with ALCL.

ELIGIBILITY:
Inclusion Criteria:

Children and adolescents with a clear diagnosis of recurrent / progressive ALCL at Shanghai Children's Medical Center or other centers since September 2017 include:

Diagnosed as ALCL, already received first-line treatment, but get disease progression; After receiving ALCL treatment has got CR then diagnosed relapse, need for pathological diagnosis.

Exclusion Criteria:

Patients with other systemic diseases, severe infections or critically illness.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2024-12 (Actual); Study Completion 2025-02 (Actual)

PRIMARY OUTCOMES:
Progression Rate | 4 weeks
  The progression rate will be obtained from the results of simple assessment after one course.
CR/CRu Rate | 8 weeks
  The CR/CRu rate will be obtained from the results of simple assessment, CT and FDG-PET after two courses.

SECONDARY OUTCOMES:
Progression-free Survival | 2 years
Overall Survival | 2 years
  Compared with historical data.

OTHER OUTCOMES:
Safety statistics: adverse reactions during the trial through NCI CTCAE version 4.0. | 2 years
  The investigators will record the adverse reactions during the trial through NCI CTCAE version 4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Yijin Gao, MD, Principal Investigator — Shanghai Children's Medical Center
Locations (1):
- Shanghai Children's Medical Center, Shanghai, Shanghai Municipality, China